CLINICAL TRIAL: NCT00224770
Title: Minimally Invasive Surgery and rtPA for Intracerebral Hemorrhage Evacuation
Acronym: MISTIE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daniel Hanley (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Genentech, Inc. (Industry); Emissary International LLC (Industry)
Responsible Party: Sponsor-Investigator, Daniel Hanley, MD, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICH01; R01NS046309 (NIH)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Medical Management (No Intervention): Standard of care medical management as per American Heart Association (AHA) guidelines.
- MISTIE Surgical Management (Active Comparator): Minimally invasive surgery (MIS) with clot lysis with recombinant tissue plasminogen activator (rt-PA).
  MIS+Cathflo Activase (drug): The intervention is a comparison of the safety and preliminary effectiveness of investigational minimally invasive surgery to place a catheter into an intracerebral hemorrhage blood clot and subsequent administration in sequential tiers of 0.3 or 1.0mg of rt-PA, CathFlo®) through the catheter once every eight hours for up to 72 hours, in addition to best medical care.
  This includes 54 intent-to-treat patients, and excludes 27 pilots.
  Interventions: Drug: MIS+Cathflo Activase (drug)
- ICES Surgical Management (Active Comparator): Intraoperative stereotactic CT-Guided Endoscopic Surgery
  Mechanical intracerebral hemorrhage removal via an endoscope utilizing the same operative-targeting arm as MISTIE arm. Best medical care was provided, but no rt-PA was administered.
  This includes 14 intent-to-treat patients, and excludes 4 pilots.
  Interventions: Procedure: Intraoperative stereotactic CT-Guided Endoscopic Surgery

INTERVENTIONS:
Drug: MIS+Cathflo Activase (drug) — MIS+Cathflo Activase (drug): The intervention is a comparison of the safety and preliminary effectiveness of investigational minimally invasive surgery to place a catheter into an intracerebral hemorrhage blood clot and subsequent administration in sequential tiers of 0.3 or 1.0mg of rt-PA, CathFlo® through the catheter once every eight hours for up to 72 hours, in addition to best medical care.
  Other Names: rtPA
  Arms: MISTIE Surgical Management
Procedure: Intraoperative stereotactic CT-Guided Endoscopic Surgery — Mechanical intracerebral hemorrhage removal via an endoscope utilizing the same operative targeting arm as MISTIE arm. No rt-PA administered, and in addition to best medical care.
  Arms: ICES Surgical Management

SUMMARY:
The purpose of this trial is to determine the safety of using a combination of minimally invasive surgery and clot lysis with rt-PA to remove intracerebral hemorrhage (ICH). The ICES arm of the trial will determine the safety of endoscopic surgery to remove ICH. All MISTIE intention to treat subjects represent the hypothesized test group. The ICES cohort is to be analyzed separately.

DETAILED DESCRIPTION:
The purpose of this trial is to determine the safety of using a combination of minimally invasive surgery and clot lysis with rt-PA to remove intracerebral hemorrhage (ICH). The procedure is to use image-based surgery (MRI or CT) to provide catheter access to ICH for the intervention, which is a one-time clot aspiration followed by instillation of rt-PA over 72 hours.

The Intraoperative stereotactic CT-guided Endoscopic Surgery (ICES) arm of the trial will determine the safety, feasibility and effectiveness of endoscopic surgery to remove ICH. This tests the first step of the MISTIE surgical procedure with an endoscope, not a rigid cannula.

We propose to test if these interventions facilitate more rapid and complete recovery of function and decreased mortality from this condition compared to conventional medical management without subjecting the patient to craniotomy. The specific objective of this trial is to test the safety of these interventions and assess their ability to remove blood clot from brain tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* GCS < 14 or a NIHSS > or equal to 6
* Spontaneous supratentorial ICH > or equal to 20cc
* Symptoms less than 12 hours prior to diagnostic CT scan (an unknown time of symptom onset is exclusionary)
* Intention to initiate surgery within 48 hours after diagnostic CT
* First dose can be given within 54 hours after diagnostic CT (delays for post surgical stabilization of catheter bleeding or because of unanticipated surgical delay are acceptable with approved waiver from the coordinating center) (Does not apply to ICES Tier)
* Six-hour clot size equal to the most previous clot size + 5 cc (as determined by an additional CT scan at least 6 hours after the initial stability scan (A*B*C)/2 method)
* SBP < 200 mmHg sustained for 6 hours recorded closest to time of randomization
* Historical Rankin score of 0 or 1
* Negative pregnancy test

Exclusion Criteria:

* Infratentorial hemorrhage (any involvement of the midbrain or lower brainstem as demonstrated by radiograph or complete third nerve palsy)
* Patients with platelet count < 100,000, INR > 1.4, or an elevated PT or APTT (reversal of coumadin is permitted but the patient must not require coumadin during the acute hospitalization). Irreversible coagulopathy either due to medical condition or prior to randomization
* Clotting disorders
* Any concurrent serious illness that would interfere with the safety assessments including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, and hematologic disease
* Patients with a mechanical valve
* Patients with unstable mass or evolving intracranial compartment syndrome
* Ruptured aneurysm, AVM, vascular anomaly
* Greater than 80 years (higher incidence of amyloid)
* Under 18 years of ag e (high incidence of occult vascular malformation)
* Pregnant (positive pregnancy test) or lactating females (likelihood of altered coagulation function associated with the high estrogen/progesterone state)
* Irreversibly impaired brainstem function (bilateral fixed, dilated pupils and extensor motor posturing), GCS less than or equal to 4
* Historical Rankin score greater than or equal to 2
* Intraventricular hemorrhage requiring external ventricular drainage
* Internal bleeding, involving retroperitoneal sites, or the gastrointestinal, genitourinary, or respiratory tracts (Does not apply to ICES Tier)
* Superficial or surface bleeding, observed mainly at vascular puncture and access sites (e.g., venous cutdowns, arterial punctures) or site of recent surgical intervention (Does not apply to ICES Tier)
* Known risk for embolization, including history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis, and subacute bacterial endocarditis (Does not apply to ICES Tier)
* In the investigator's opinion, the patient is unstable and would benefit from a specific intervention rather than supportive care plus or minus MIS+rtPA
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous trial of ICH treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2005-08; Primary Completion 2012-08 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F. Hanley, MD, Study Chair — Johns Hopkins University; Mario Zuccarello, MD, Principal Investigator — University of Cincinnati; Paul Vespa, MD, Principal Investigator — University of California, Los Angeles
Locations (29):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurosurgical Associates, Phoenix, Arizona
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, San Diego, San Diego, California
  - Hartford Hospital, Hartford, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - University of Maryland Medical Systems, Baltimore, Maryland
  - Johns Hopkins University/Bayview Medical Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - JFK Medical Center New Jersey, Edison, New Jersey
  - Mt. Sinai Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western University, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas, Houston, Houston, Texas
  - University of Texas HSC, San Antonio, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Montreal Neurological Institute at McGill University, Montreal, Quebec, Canada
- University of Heidelberg, Heidelberg, Germany
- Newcastle General Hospital, Newcastle, United Kingdom

REFERENCES:
- [Derived] Hansen BM, Ullman N, Muschelli J, Norrving B, Dlugash R, Avadhani R, Awad I, Zuccarello M, Ziai WC, Hanley DF, Thompson RE, Lindgren A; MISTIE and CLEAR Investigators. Relationship of White Matter Lesions with Intracerebral Hemorrhage Expansion and Functional Outcome: MISTIE II and CLEAR III. Neurocrit Care. 2020 Oct;33(2):516-524. doi: 10.1007/s12028-020-00916-4. PMID 32026447
- [Derived] Vespa P, Hanley D, Betz J, Hoffer A, Engh J, Carter R, Nakaji P, Ogilvy C, Jallo J, Selman W, Bistran-Hall A, Lane K, McBee N, Saver J, Thompson RE, Martin N; ICES Investigators. ICES (Intraoperative Stereotactic Computed Tomography-Guided Endoscopic Surgery) for Brain Hemorrhage: A Multicenter Randomized Controlled Trial. Stroke. 2016 Nov;47(11):2749-2755. doi: 10.1161/STROKEAHA.116.013837. Epub 2016 Oct 6. PMID 27758940
- [Derived] Hanley DF, Thompson RE, Muschelli J, Rosenblum M, McBee N, Lane K, Bistran-Hall AJ, Mayo SW, Keyl P, Gandhi D, Morgan TC, Ullman N, Mould WA, Carhuapoma JR, Kase C, Ziai W, Thompson CB, Yenokyan G, Huang E, Broaddus WC, Graham RS, Aldrich EF, Dodd R, Wijman C, Caron JL, Huang J, Camarata P, Mendelow AD, Gregson B, Janis S, Vespa P, Martin N, Awad I, Zuccarello M; MISTIE Investigators. Safety and efficacy of minimally invasive surgery plus alteplase in intracerebral haemorrhage evacuation (MISTIE): a randomised, controlled, open-label, phase 2 trial. Lancet Neurol. 2016 Nov;15(12):1228-1237. doi: 10.1016/S1474-4422(16)30234-4. Epub 2016 Oct 11. PMID 27751554
- [Derived] Muschelli J, Ullman NL, Sweeney EM, Eloyan A, Martin N, Vespa P, Hanley DF, Crainiceanu CM. Quantitative Intracerebral Hemorrhage Localization. Stroke. 2015 Nov;46(11):3270-3. doi: 10.1161/STROKEAHA.115.010369. Epub 2015 Oct 8. PMID 26451031
- [Derived] Webb AJ, Ullman NL, Morgan TC, Muschelli J, Kornbluth J, Awad IA, Mayo S, Rosenblum M, Ziai W, Zuccarrello M, Aldrich F, John S, Harnof S, Lopez G, Broaddus WC, Wijman C, Vespa P, Bullock R, Haines SJ, Cruz-Flores S, Tuhrim S, Hill MD, Narayan R, Hanley DF; MISTIE and CLEAR Investigators. Accuracy of the ABC/2 Score for Intracerebral Hemorrhage: Systematic Review and Analysis of MISTIE, CLEAR-IVH, and CLEAR III. Stroke. 2015 Sep;46(9):2470-6. doi: 10.1161/STROKEAHA.114.007343. Epub 2015 Aug 4. PMID 26243227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 110 patients were randomized to the trial, and 31 were recruited as pilot patients.
Pre-assignment Details: Each study center was required to demonstrate proficiency in the technical aspects of enrollment, stabilization, surgery, and drug administration. This proficiency was demonstrated on at least one pilot patient prior to randomization of the first patient in the investigational cohort of 110 randomized patients.
Groups:
- MISTIE Surgical Management: Minimally invasive surgery (MIS) with clot lysis with recombinant tissue plasminogen activator (rt-PA).
  MIS+Cathflo Activase (drug): The intervention is a comparison of the safety and preliminary effectiveness of investigational minimally invasive surgery to place a catheter into an intracerebral hemorrhage blood clot and subsequent administration in sequential tiers of 0.3 or 1.0mg of rt-PA, CathFlo® through the catheter once every eight hours for up to 72 hours, in addition to best medical care.
  This includes 54 intent-to-treat patients, and excludes 27 pilots.
- ICES Surgical Management: Intraoperative stereotactic CT-Guided Endoscopic Surgery (ICES)
  Mechanical intracerebral hemorrhage removal via an endoscope utilizing the same operative-targeting arm as MISTIE arm. Best medical care was provided, but no rt-PA was administered.
  This includes 14 intent-to-treat patients, and excludes 4 pilots.
Period: Overall Study
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Started | 42 | 54 | 14
Completed | 38 | 52 | 14
Not Completed | 4 | 2 | 0
Not completed — Lost to Follow-up | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The decision was made to exclude the pilot patients from the analysis...
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management | Total
Number analyzed (Participants) | 42 | 54 | 14 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 25 | 9 | 52
  >=65 years | 24 | 29 | 5 | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [49.5 to 73] | 60 [54 to 69] | 59 [53.2 to 68.2] | 61 [53.3 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 5 | 38
  Male | 28 | 35 | 9 | 72
Region of Enrollment [Number; unit: participants]
  United States | 41 | 53 | 14 | 108
  United Kingdom | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety Outcome Number 1: Rate of Mortality
Description: Percentage of participants who died during the first 30 days after randomization.
Time Frame: 30 days from randomization
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Number analyzed (Participants) | 42 | 54 | 14
percentage of participants | 9.5 [3.3 to 20.5] | 14.8 [7.6 to 25.1] | 7.1 [0.4 to 29.7]
Statistical Analysis 1: Comparison: Medical Management vs MISTIE Surgical Management; Null hypothesis is that rate of mortality within 30 days is the same between the two groups. The alternative hypothesis tests whether MISTIE surgical management has a higher rate of mortality than the medical arm; Test type: Superiority or Other; p = 0.324, Fisher Exact; One-sided test; Risk Difference (RD) = 5.3, 95% CI 1-sided [upper limit 16.2], Standard Error of Mean 6.6 — MISTIE rate=14.8, 95% upper limit=25.1; medical rate=9.5, 95% upper limit=20.5; comparison considers MISTIE rate minus medical rate
Statistical Analysis 2: Comparison: Medical Management vs ICES Surgical Management; Null hypothesis is that rate of mortality within 30 days is the same between the two groups. The alternative hypothesis tests whether ICES surgical management has a higher rate of mortality than the medical arm; Test type: Superiority or Other; p = 0.633, Fisher Exact; One-sided test; Risk Difference (RD) = -2.4, 95% CI 1-sided [upper limit 11.2], Standard Error of Mean 8.2 — ICES rate=7.1, 95% upper limit=29.7; medical rate=9.5, 95% upper limit=20.5; comparison considers ICES rate minus medical rate

2. Primary Outcome: Safety Outcome Number 2: Rate of Procedure-related Mortality
Description: Percentage of participants who died during the first 7 days after randomization.
Time Frame: 7 days from randomization
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Number analyzed (Participants) | 42 | 54 | 14
percentage of participants | 0 [0 to 6.9] | 5.6 [1.5 to 13.7] | 0 [0 to 19.3]
Statistical Analysis 1: Comparison: Medical Management vs MISTIE Surgical Management; Null hypothesis is that rate of procedure-related mortality within 7 days is the same between the two groups. The alternative hypothesis tests whether MISTIE surgical management has a higher rate of procedure-related mortality than the medical arm; Test type: Superiority or Other; p = 0.174, Fisher Exact; One-sided test; Risk Difference (RD) = 5.6, 95% CI 1-sided [upper limit 11.7], Standard Error of Mean 3.1 — MISTIE rate=5.6, 95% upper limit=13.7; medical rate=0.0, 95% upper limit=6.9; comparison considers MISTIE rate minus medical rate

3. Primary Outcome: Safety Outcome Number 3: Rate of Cerebritis, Meningitis, Bacterial Ventriculitis
Description: Percentage of participants who had a bacterial brain infection (cerebritis, meningitis, ventriculitis) within 30 days of randomization.
Time Frame: 30 days from randomization
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Number analyzed (Participants) | 42 | 54 | 14
percentage of participants | 2.4 [0.1 to 10.8] | 0 [0 to 5.4] | 0 [0 to 19.3]
Statistical Analysis 1: Comparison: Medical Management vs MISTIE Surgical Management; Null hypothesis is that rate of cerebritis, meningitis and ventriculitis within 30 days is the same between the two groups. The alternative hypothesis tests whether MISTIE surgical management has a higher rate of these infections than medical; Test type: Superiority or Other; p = 0.437, Fisher Exact; One-sided test; Risk Difference (RD) = -2.4, 95% CI 1-sided [upper limit 1.5], Standard Error of Mean 2.4 — MISTIE rate=0.0, 95% upper limit=5.4; medical rate=2.4, 95% upper limit=10.8; comparison considers MISTIE rate minus medical rate
Statistical Analysis 2: Comparison: Medical Management vs ICES Surgical Management; Null hypothesis is that rate of cerebritis, meningitis and ventriculitis within 30 days is the same between the two groups. The alternative hypothesis tests whether ICES surgical management has a higher rate of these infections than medical; Test type: Superiority or Other; p = 0.750, Fisher Exact; One-sided test; Risk Difference (RD) = -2.4, 95% CI 1-sided [upper limit 1.5], Standard Error of Mean 2.4 — ICES rate=0.0, 95% upper limit=19.3; medical rate=2.4, 95% upper limit=10.8; comparison considers ICES rate minus medical rate

4. Primary Outcome: Safety Outcome Number 4: Rate of Symptomatic Rebleeding
Description: The difference in the rate of symptomatic rebleeding 72 hours post last dose.
Time Frame: 72 hours post last dose
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- ICES Surgical Management: Intraoperative stereotactic CT-Guided Endoscopic Surgery (ICES)
  Mechanical intracerebral hemorrhage removal via an endoscope utilizing the same operative targeting technique as the MISTIE arm. No rt-PA administered, and in addition to best medical care.
  This includes 14 intent-to-treat patients, and excludes 4 pilots.
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Number analyzed (Participants) | 42 | 54 | 14
percentage of participants | 2.4 [0.1 to 10.8] | 5.6 [1.5 to 13.7] | 0 [0 to 19.3]
Statistical Analysis 1: Comparison: Medical Management vs MISTIE Surgical Management; Null hypothesis is that rate of symptomatic rebleeding 72 hours post last dose is the same between the two groups. The alternative hypothesis tests whether MISTIE surgical management has a higher rate of symptomatic rebleeding than the medical arm; Test type: Superiority or Other; p = 0.409, Fisher Exact; One-sided test; Risk Difference (RD) = 3.2, 95% CI 1-sided [upper limit 9.6], Standard Error of Mean 3.9 — MISTIE rate=5.6, 95% upper limit=13.7; medical rate=2.4, 95% upper limit=10.8; comparison considers MISTIE rate minus medical rate
Statistical Analysis 2: Comparison: Medical Management vs ICES Surgical Management; Null hypothesis is that rate of symptomatic rebleeding 72 hours post last dose is the same between the two groups. The alternative hypothesis tests whether ICES surgical management has a higher rate of symptomatic rebleeding than the medical arm; Test type: Superiority or Other; p = 0.750, Fisher Exact; One-sided test; Risk Difference (RD) = -2.4, 95% CI 1-sided [upper limit 2.2], Standard Error of Mean 2.4 — [estimate comment as in outcome 3, analysis 2]

5. Secondary Outcome: Ordinal Modified Rankin Scale (mRS) at Day 180
Description: Ordinal distribution of the Modified Rankin Scale score at 180 days. The mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale ranges from 0-6: (0) no symptoms at all, (1) no significant disability despite symptoms; able to carry out all usual duties and activities, (2) slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance, (3) moderate disability; requiring some help, but able to walk without assistance, (4) moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance, (5) severe disability; bedridden, incontinent and requiring constant nursing care and attention, (6) dead.
Time Frame: 180 days from randomization
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Number analyzed (Participants) | 38 | 52 | 14
units on a scale | 4 [4 to 6] | 4 [3 to 6] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Medical Management vs MISTIE Surgical Management; Null hypothesis is that the distributions of the mRS values for both groups are the same. The alternative hypothesis is that the distributions are not the same; Test type: Superiority or Other; p = 0.468, Wilcoxon (Mann-Whitney); Two-sided test
Statistical Analysis 2: Comparison: Medical Management vs ICES Surgical Management; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.294, Wilcoxon (Mann-Whitney); Two-sided test

6. Secondary Outcome: Ordinal Modified Rankin Scale (mRS) at Day 365
Description: Ordinal distribution of the Modified Rankin Scale score at 365 days. The mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale ranges from 0-6: (0) no symptoms at all, (1) no significant disability despite symptoms; able to carry out all usual duties and activities, (2) slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance, (3) moderate disability; requiring some help, but able to walk without assistance, (4) moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance, (5) severe disability; bedridden, incontinent and requiring constant nursing care and attention, (6) dead.
Time Frame: 365 days from randomization
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Number analyzed (Participants) | 24 | 20 | 12
units on a scale | 4.5 [3.5 to 6] | 4 [2 to 6] | 3.5 [3 to 5]
Statistical Analysis 1: Comparison: Medical Management vs MISTIE Surgical Management; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.395, Wilcoxon (Mann-Whitney); Two-sided test
Statistical Analysis 2: Comparison: Medical Management vs ICES Surgical Management; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.175, Wilcoxon (Mann-Whitney); Two-sided test

7. Secondary Outcome: Clot Size Reduction by End of Treatment
Description: The percentage of blood clot resolved by the end of treatment CT scan compared to the stability CT scan.
Time Frame: Time from randomization until end of treatment, up to 10 days
Measure: Median (Inter-Quartile Range); unit: percentage of blood clot resolved
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Number analyzed (Participants) | 42 | 54 | 14
percentage of blood clot resolved | 3.9 [-0.06 to 10.2] | 64.3 [43.3 to 74.1] | 69.5 [59.0 to 86.0]
Statistical Analysis 1: Comparison: Medical Management vs MISTIE Surgical Management; Null hypothesis is that the distributions of percentage of blood clot resolved are the same between the two groups. The alternative hypothesis is that the distributions are not the same; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Two-sided test
Statistical Analysis 2: Comparison: Medical Management vs ICES Surgical Management; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Two-sided test

8. Secondary Outcome: Post-operative Clot Size Reduction
Description: The percentage of blood clot resolved by the end of treatment CT scan compared to the post-operative CT scan for surgical patients.
Time Frame: Time from post-operation until end of treatment, up to 10 days
Population: Analysis population only includes surgical patients.
Measure: Median (Inter-Quartile Range); unit: percentage of blood clot resolved
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Number analyzed (Participants) | 0 | 54 | 14
percentage of blood clot resolved |  | 56.7 [23.6 to 68.4] | -6.4 [-21.3 to 4.0]
Statistical Analysis 1: Comparison: MISTIE Surgical Management; Null hypothesis is that the median percent resolved is 0. The alternative hypothesis is that the median percent resolved is not equal to 0; Test type: Superiority or Other; p < 0.0001, Sign test; Two-sided test
Statistical Analysis 2: Comparison: ICES Surgical Management; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.791, Sign test; Two-sided

9. Primary Outcome: Efficacy Outcome Number 1: Dichotomized Modified Rankin Scale (mRS) at Day 180
Description: Percentage of participants with dichotomized mRS score in 0-3 range. The mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale ranges from 0-6: (0) no symptoms at all, (1) no significant disability despite symptoms; able to carry out all usual duties and activities, (2) slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance, (3) moderate disability; requiring some help, but able to walk without assistance, (4) moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance, (5) severe disability; bedridden, incontinent and requiring constant nursing care and attention, (6) dead
Time Frame: 180 days from randomization
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Number analyzed (Participants) | 38 | 52 | 14
percentage of participants | 23.7 [12.9 to 37.7] | 34.6 [23.7 to 46.9] | 42.9 [20.6 to 67.5]
Statistical Analysis 1: Comparison: Medical Management vs MISTIE Surgical Management; Null hypothesis is that the proportion with mRS score of 0-3 at 180 days is the same between the two groups. The alternative hypothesis tests whether MISTIE surgical management has a higher proportion than the medical arm; Test type: Superiority or Other; p = 0.189, Fisher Exact; One-sided test; Risk Difference (RD) = 10.9, 95% CI 1-sided [upper limit 26.6], Standard Error of Mean 9.5 — MISTIE rate=34.6, 95% upper limit=46.9; medical rate=23.7, 95% upper limit=37.7; comparison considers MISTIE rate minus medical rate
Statistical Analysis 2: Comparison: Medical Management vs ICES Surgical Management; Null hypothesis is that the proportion with mRS score of 0-3 at 180 days is the same between the two groups. The alternative hypothesis tests whether ICES surgical management has a higher proportion than the medical arm; Test type: Superiority or Other; p = 0.156, Fisher Exact; One-sided test; Risk Difference (RD) = 19.2, 95% CI 1-sided [upper limit 43.7], Standard Error of Mean 14.9 — ICES rate=42.9, 95% upper limit=67.5; medical rate=23.7, 95% upper limit=37.7; comparison considers ICES rate minus medical rate

ADVERSE EVENTS:
Arm/Group | Medical Management | MISTIE Surgical Management | ICES Surgical Management
Serious Adverse Events (participants affected / at risk) | 23/42 | 28/54 | 6/14
Other Adverse Events (participants affected / at risk) | 24/42 | 41/54 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Management (N=42) | MISTIE Surgical Management (N=54) | ICES Surgical Management (N=14)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage: Tissue, Enlargement (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Intracranial hemorrhage: Tissue, New (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Intracranial hemorrhage: Ventricular system, New (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial hypertension (Nervous system disorders) | 4 (4) | 2 (3) | 0 (0)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 4 (4) | 3 (3) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Left renal mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PVC's, bigemeny (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Anoxic brain injury (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitits (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 1 (1)
Pulmonary embolism (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 0 (0)
Seizure (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 3 (5) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ventilatory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage: Catheter Tract, New (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage: Catheter Tract, Enlargement (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage: Ventricular system, Enlargement (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Herniation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Management (N=42) | MISTIE Surgical Management (N=54) | ICES Surgical Management (N=14)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Fever (General disorders) | 6 (6) | 13 (14) | 3 (3)
Hematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 6 (6) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 0 (0)
Lung infection (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (2) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6) | 2 (2)
Seizure (Nervous system disorders) | 3 (5) | 4 (4) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 5 (5) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 9 (9) | 0 (0)
Ventilatory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 8 (11) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (6) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 3 (5) | 0 (0)
Intracranial hemorrhage: Catheter Tract, Enlargement (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
Intracranial hemorrhage: Catheter Tract, New (Nervous system disorders) | 0 (0) | 6 (6) | 0 (0)
Intracranial hemorrhage: Tissue, Enlargement (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
Intracranial hemorrhage: Ventricular system, Enlargement (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Localized edema (General disorders) | 0 (0) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 0 (0)
HCAP (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound reclosure after serious fluid leak (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the funding agency (NIH/NINDS) can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the funding agency for review. The funding agency cannot require changes to the communication and cannot extend the embargo.